CLINICAL TRIAL: NCT05768386
Title: A Long-Term Follow-Up Study in Subjects With Severe Hemophilia A Who Received BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in a Prior BioMarin Clinical Trial
Brief Title: A Long-Term Follow-Up Study in Severe Hemophilia A Subjects Who Received BMN 270 in a Prior BioMarin Clinical Trial (270-401)
Acronym: GENEr8-LTE
Status: Enrolling by invitation | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 270-401; 2022-001246-38 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
Keywords: Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases; Inborn; Factor VIII; Coagulants
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BMN 270 clinical development program consists of multiple interventional studies designed to assess the safety and efficacy of a single infusion of BMN 270 for at least 5 years post-infusion. This long-term follow-up study is needed to help further understand the long-term safety of BMN 270 beyond 5 years and to assess the durability of efficacy.

DETAILED DESCRIPTION:
Study 270-401 will collect additional follow-up data in a single study for approximately 10 years among all subjects who consent to participate and have completed their primary treatment study (ie, for any study in which they received BMN 270).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed their primary treatment study or be currently enrolled in the primary treatment study at the time of closure by the Sponsor. Participants may enroll in 270-401 even if they have restarted FVIII prophylaxis or other hemophilia A treatment.
* Subjects must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. If the subject is unable to provide consent, a legally authorized representative may provide written informed consent.

Exclusion Criteria:

* Participants who do not directly enroll in 270-401 at the time of the study completion visit in their primary treatment study should enroll in 270-401 within 4 months of the date of that study completion visit. If a participant wishes to enroll in 270-401 after 4 months, they must receive prior approval from the Medical Monitor.
* Participants must be overtly healthy and not have any condition that, in the opinion of the Investigator or Medical Monitor, would prevent the participant from fully complying with the requirements of the study and/or would impact or interfere with evaluation and interpretation of the study data (including, if applicable, advanced HIV disease).
* Where applicable, per country regulation, the participant must not currently be committed to an institution by virtue of an order issued either by judicial or administrative authorities.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subjects must have completed their primary treatment study in which they were dosed BMN 270. Subjects may enroll in 270-401 even if they have restarted FVIII prophylaxis or other hemophilia A treatment.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long-term safety of BMN 270 | Duration of study (10 years)
  Occurrence of adverse drug reactions, serious adverse events, and events of special interest.

SECONDARY OUTCOMES:
Evaluate the long-term effects of BMN 270 in subjects with hemophilia A previously treated in a BioMarin clinical trial | Duration of study (10 years)
  Changes in annualized bleeding rate (ABR) (treated bleeds and all bleeds) and FVIII activity measured over time (CSA and OSA)
Evaluate the use of hemostatic agents (ie, emicizumab) | Duration of study (10 years)
  Annualized use of concomitant hemostatic medications (annualized FVIII utilization and annualized FVIII infusion rate)
Evaluate the long-term impact of BMN 270 on HRQoL | Duration of study (10 years)
  Changes in Haemo-QOL-A

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (41):
- United States (13):
  - Orthopedic Institute for Children, Orthopedic Hemophilia Treatment Center, Los Angeles, California
  - UC Davis Hemophilia Treatment Center, Sacramento, California
  - University of California San Diego, Hemophilia & Thrombosis Treatment Center, San Diego, California
  - University of California San Francisco - Moffit Hospital, Outpatient Hematology Clinic, San Francisco, California
  - UCN Hemophilia and Thrombosis Center, Shandon, California
  - Hemophilia and Thrombosis Center at the University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - St Joseph's Children's Hospital, Center for Bleeding and Clotting Disorders, Tampa, Florida
  - University Medical Center, Inc,; DBA University of Louisville Hospital, James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Michigan, Pediatric Hematology and Oncology, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Hemophilia and Thrombosis Center, Detroit, Michigan
  - Washington University School of Medicine, Department of Pediatrics, Division of Hematology/Oncology, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
- Australia (5):
  - Royal Prince Alfred Hospital, Institute of Haematology, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- University Hospitals Leuven, Campus Gasthuisberg, Department of Heart and Vascular Disease, Leuven, Belgium
- Brazil (4):
  - Holy Spirit Hematology and Hemotherapy Center, Vitória, Espírito Santo
  - Arthur De Siqueira Cavalcanti Hematology State Institute / Coordinating Hemocenter, Rio de Janeiro, Rio de Janeiro
  - Campinas University Clinical Hospital, Hematology and Hemotherapy Center (Hemocentro UNICAMP), Campinas, São Paulo
  - Sao Paulo University Clinical Hospital, São Paulo, São Paulo
- France (2):
  - CHRU Lille Hospital Center Heart-Lung Institute, Lille
  - CHU La Timone - La Timone Children's Hospital, Marseille
- Germany (2):
  - University Hospital Bonn, Institute of Experimental Hematology and Transfusion Medicine, Hemophilia Care Center, Bonn, North Rhine-Westphalia
  - Vivantes Hospital in Friedrichshain, Berlin, State of Berlin
- Chaim Sheba Medical Center, National Institute of Hemophilia and Coagulation, Ramat Gan, Israel
- Maggiore Polyclinic Hospital, Foundation IRCCS Ca' Granda, Center for Hemophilia and Thrombosis "Angelo Bianchi Bonomi", Milan, Italy
- Charlotte Maxeke Johannesburg Academic Hospital, Hemophilia Comprehensive Care Center, Johannesburg, South Africa
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea
- Spain (2):
  - University Hospital Virgen del Rocio (HUVR), Hematology Pediatrics, Seville, Andalusia
  - Hospital Teresa Herrera, Department of Hematology and Hemotherapy, Unit of Hemostasis and Thrombosis, A Coruña, Galicia
- United Kingdom (8):
  - Addenbrooke's Hospital, Hemophilia and Thrombophilia Center, Cambridge
  - Glasgow Royal Infirmary, Department of Hematology, Glasgow
  - Hammersmith Hospital, Clinical Research Facility, Centre for Translational and Experimental Medicine, London
  - Queen Elizabeth Hospital Birmingham. Adult Hemophilia Centre, West Midlands Adult Comprehensive Care Hemophilia Centre, London
  - Royal London Hospital, Barts and the London Hemophilia Center, London
  - St Thomas' Hospital, Centre for Hemophilia, Hemostasis and Thrombosis, London
  - Nuffield Orthopaedic Centre, Hemophilia & Thrombosis Center, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton